CLINICAL TRIAL: NCT00274066
Title: The Acute Bronchodilator Effects of a Single Dose (2 Puffs) of the Shortacting Anticholinergic Ipratropium Bromide (40μg) and the Short-acting Beta-adrenergic Fenoterol (200μg) in Comparison to Placebo on Top of Pharmacodynamic Steady State of Once Daily Tiotropium (18μg) Inhalation Capsule in Patients With Chronic Pulmonary Disease (COPD)
Brief Title: Acute Bronchodilator Response of a Single Dose of Atrovent or Berotec on Top of Pharmacodynamic Steady State of Spiriva
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.258
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Ipratropium; Fenoterol

INTERVENTIONS:
Drug: Tiotropium + placebo
Drug: Tiotropium + ipratropium
Drug: Tiotropium + fenoterol

SUMMARY:
To evaluate acute effect of single dose of ipratropium (Atrovent) or fenoterol (Berotec) in comparison to placebo when given to COPD patients on pharmacodynamic steady state of tiotropium (Spiriva)

DETAILED DESCRIPTION:
In case mono-bronchodilator therapy does not control symptoms of COPD adequately or if regular maintenance therapy is desired, a therapeutic intervention with a combination of bronchodilators is recommended. The risks of side-effects increases with increasing dose of any drug and, therefore, the most important rationale for combination therapy is a very favourable ratio of efficacy and safety. Knowing that anticholinergic and beta-adrenergic agents achieve their bronchodilating effects by different mechanisms, in particular the combination of these agents has proven to be beneficial in the management of COPD. Based on the established clinical benefits, tiotropium is an attractive and promising agent for the first-line long-term maintenance therapy in COPD. This also implies that a therapeutic intervention with other bronchodilators will be prescribed in daily practice. At present no studies on combination therapy with short-acting agents are available. Therefore, using a double-blind, randomised, crossover design, the bronchodilator effects of single doses of ipratropium or fenoterol were compared with placebo when added on top of steady state tiotropium. Patients were pre-treated with tiotropium to achieve this pharmacodynamic steady state. Serial lung function tests (FEV1, FVC, Raw, sGaw) were conducted following add-on of the short-acting bronchodilators or placebo.

Study Hypothesis:

H0: there is no difference between treatments in mean peak FEV1 H1: there is a difference between treatments in mean peak FEV1

Comparison(s):

Add-on of placebo was compared to add-on of ipratropium or add-on of fenoterol. The comparison of ipratropium with placebo was primary. The other 2 pair-wise comparisons were secondary.

ELIGIBILITY:
Inclusion:

* diagnosis of COPD
* FEV1 < 60% of predicted
* FEV1 < 70% of FVC
* smoking history of 10 pack-years

Exclusion:

* significant other disease than COPD
* history of asthma, allergic rhinitis or blood eosinophil count > 600mm3
* cardiac arrhythmia requiring drug therapy
* symptomatic prostatic hypertrophy, bladder neck obstruction or narrow-angle glaucoma
* recent history of MI (within past year)
* history of cancer within past 5 years
* life-threatening pulmonary obstruction
* cystic fibrosis or bronchiectasis; tuberculosis
* pulmonary resection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2002-10; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Peak FEV1 response, defined as the peak FEV1 minus the steady-state baseline FEV | up to 37 days

SECONDARY OUTCOMES:
Peak FVC response in the six-hour observation period following administration of the first single dose of randomised treatment | up to 37 days
FEV1 and FVC response one hour after the second dose of randomised treatment | up to 37 days
Individual FEV1 and FVC measurements at each time point | up to 37 days
sGaw and Raw measured at 1 and 6 hour after the first dose of randomised treatment and at 1 hour after the second dose of randomised treatment | up to 37 days
All adverse events | up to 37 days
Pulse rate | up to 37 days
Sitting blood pressure in conjunction with spirometry | up to 37 days
ECG recorded one hour after the first dose of randomised treatment | up to 37 days
Physical examination at baseline (Visit 1) and at the conclusion of patient participation in the trial | up to 37 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim BV/Alkmaar
Locations (5):
- Netherlands (5):
  - Twenteborg Ziekenhuis, Almelo
  - Amphia Ziekenhuis, Breda
  - Boehringer Ingelheim Investigational Site, Groningen
  - Afdeling longziekten, Winschoten
  - Gelre Ziekenhuizen, Zutphen

REFERENCES:
- [Derived] Kerstjens HA, Bantje TA, Luursema PB, Sinninghe Damste HE, de Jong JW, Lee A, Wijker SP, Cornelissen PJ. Effects of short-acting bronchodilators added to maintenance tiotropium therapy. Chest. 2007 Nov;132(5):1493-9. doi: 10.1378/chest.06-3059. Epub 2007 Sep 21. PMID 17890476